CLINICAL TRIAL: NCT04199663
Title: Secondary Prevention Treatments and Activities Post Myocardial Infarction Underlying the Risk of Recurrent Hard Cardiovascular Outcomes Associated With Socioeconomic Status
Brief Title: Socioeconomic Status, Secondary Prevention Activities and Recurrence After a Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Per Svensson, Associate professor, Karolinska Institutet
Other Study IDs: 3
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Socioeconomic Status; Secondary Prevention; Myocardial Infarction; Cardiovascular Disease; Stroke
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 88 Months

GROUPS / COHORTS (1):
- categories of Socioeconomic Status (SES): by proxy gender- and calendar year-specific quintiles of disposable income per household consumption unit.
  In logistic regression models of associations with secondary prevention activities and established treatment goals: highest vs. lowest income quintile.
  In multivariable Cox regression analyses with stepwise built models: quintiles of disposable income and models including covariates level of education and marital status.

SUMMARY:
This is a nationwide cohort study on real-world patients (n≈30,000) surviving a first myocardial infarction (MI) 2006-2013 and alive to attend a routine 1-year follow-up. Associations between Socioeconomic Status (SES) and secondary preventive actions (SPAs) throughout the first year is studied and assessed as possible mechanisms underlying the increased risk of a first recurrent hard cardiocvascular (CV) outcome, recurrent atherosclerotic cardiovascular disease (rASCVD), in patients with low Socioeconomic Status during long-term follow-up (2006-2018).

ELIGIBILITY:
Inclusion Criteria:

* Swedish resident
* Alive and registered in The Swedish Websystem for Enhancement and Development of Evidence based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART)'s secondary prevention subregistry between 1 January 2006 and 31 December 2013 at the 1-year-revisit

Exclusion Criteria:

* Age >76 years at baseline
* Missing data for disposable household income
* History of MI, stroke, coronary artery bypass graft (CABG), or percutaneous coronary intervention (PCI) prior to the index MI
* Not present in initial care registry (RiksHIA)
* Date of index MI before 2004 or missing
* revisit outside 13±2 month window post-MI

Ages: 18 Years to 76 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: large nation-wide population of consecutive patients with assumed stable coronary heart disease after a myocardial infarction (first manifestation of atherosclerotic cardiovascular disease) in a tax-funded health care system.
Sampling Method: Probability Sample
Enrollment: 30191 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
first recurrent atherosclerotic cardiovascular disease event (rASCVD) | from date of 1-year visit post-MI (baseline) until date of outcome, censoring or study end (2018)
  composite outcome including non-fatal MI (I210-I214, I219, I220, I221, I228 or I229) or coronary heart disease death (CHD) (I210-I214, I219, I220, I221, I228, I229, I461 or I469) or fatal or non-fatal ischemic stroke (I630-I635, I638 or I639) according to the International Classification of Diseases 10th edition (ICD-10)

OTHER OUTCOMES:
Goal: physical training program | at 1-year revisit
  participated in organized physical training program after the initial care
Goal: LDL-C goal | at 1-year revisit
  attained LDL-C level below treatment target
Goal: Blood pressure goal | at 1-year revisit
  attained blood pressure levels below treatment target
Goal: smoking cessation | at 1-year revisit
  Patients being current smokers at their initial care who successfully quit smoking.
Goal: physical activity | at 1-year revisit
  reported >30 minutes of physical activity ≥5 times a week
Goal: statin treatment | at 1-year revisit
  on statin treatment 1 year after the index MI
Goal: Renin-angiotensin-aldosteron system (RAAS)-inhibition | at 1-year revisit
  Patients with congestive heart failure, diabetes or hypertension at the index Mi on treatment with angiotensin converting enzyme inhibitor or angiotensin receptor blocker.
Goal: HbA1c goal | at 1-year revisit
  Patients with diabetes with attained HbA1c treatment target
SPA: cardiac rehabilitation program | during 1st year after initial care
  participation in structured program after the index MI
SPA: diet course | during 1st year after initial care
  participation in course after the index MI
SPA: statin intensity increase | 2 months or 1 year after initial care
  statin intensity increase decided at routine revisits (Dosages categorized into high (Rosuvastatin 20-40 mg or Atorvastatin 40-80 mg), moderate (Rosuvastatin 5-10 mg, Atorvastatin 10-20 mg, or Simvastatin 20-40 mg) and low (Simvastatin 10 mg))
SPA: high intensity statins | at 1-year revisit
  on high intensity statin treatment (Rosuvastatin 20-40 mg or Atorvastatin 40-80 mg)
SPA: LDL-C reduction | 2 months and 1 year after initial care
  LDL-C reduction between routine revisits
SPA: lipid monitoring | 2 months or 1 year after initial care
  Blood lipid panel measured
SPA: type of follow-up | 2 month revisit
  decided follow-up by office revisit or by phone
SPA: reperfusion | initial care
  type of reperfusion treatment chosen in STEMI and NSTEMI
SPA: revascularized | initial care
  achieved complete revascularization in STEMI and NSTEMI
SPA: staged procedure | initial care
  Decision on continued invasive procedures at a later stage
SPA: smoking cessation counseling | 2 months or 1 year after initial care
  received through cessation program or counseling
SPA: HbA1c monitoring | during initial care, at 2 months and 1 year after initial care
  Patients with diabetes at initial care having their HbA1c measured at least twice
SPA: Anti-stress program | 1 year after initial care
  Patients reporting anxiety or sadness participating in anti-stress program
SPA: counter-metabolic syndrome actions | 2 months or 1 year after initial care
  Patients with the metabolic syndrome participating in physical training and diet course or in cardiac rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Per O Svensson, MD PhD, Principal Investigator — Department of Clinical Science and Education, Söderjukhuset